CLINICAL TRIAL: NCT05590221
Title: Study to Evaluate the Efficacy and Safety of Relmacabtagene Autoleucel (Relma-cel) as First-Line Therapy in Adult Participants With High-Risk Large B-Cell Lymphoma
Brief Title: Relmacabtagene Autoleucel as First-Line Therapy for High-Risk Large B-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029011
Record Dates: First submitted 2022-10-12; First posted 2022-10-21 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-11

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — relmacabtagene autoleucel; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relmacabtagene Autoleucel (Experimental): Participants will receive cyclophosphamide250 mg/m^2/day intravenously (IV) and fludarabine 25 mg/m^2/day IV conditioning chemotherapy for 3 days followed by Relmacabtagene Autoleucel administered as a single IV infusion at a target dose of 1 x 10^8 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells on Day 1.
  Interventions: Biological: Relmacabtagene Autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Relmacabtagene Autoleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: JWCAR029
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert

SUMMARY:
The primary objective of this study is to estimate the efficacy of Relmacabtagene Autoleucel in participants with high-risk large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, single-arm trial, assessed the efficacy and safety of JWCAR029(relma-cel) as part of first-line therapy after an incomplete first-line treatment regimen of two cycles of chemoimmunotherapy. High-risk LBCL was defined by the dynamic risk assessment of interim PET2+, together with either double- or triple-hit lymphomas or high-intermediate- and high-risk IPI scores (≥3). All sujects will be followed for 2 years following JWCAR029 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old;
2. Sign on the informed consent;
3. Histologically confirmed large B-cell lymphoma that also meets the definition of high-risk large B-cell lymphoma as a lymphoma International Prognostic Index (IPI) score of 3-5 and/or high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement (double/triple-hit lymphoma) (DHL/THL) and must be treated with 2 cycles of CD20 monoclonal antibodies combined with anthracyclines. Presence of positive PET assessable lesions (DS score of 4 or 5) as determined by the Lugano criteria (Cheson et al., 2014)；
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Expected survival greater than 12 weeks；
6. Adequate organ function：

   1. Absolute neutrophil count ≥ 1000/μL；Absolute lymphocyte count ≥ 100/μL； Platelet count ≥ 75,000/μL；Hb ≥ 80g/L；
   2. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (Cockcroft-Gault formula) > 50 mL/min (serum creatinine clearance due to lymphoma mass compression should be > 30 mL/min)；
   3. Serum alanine aminotransferase (ALT) ≤ 5 upper limit of normal (ULN) and total bilirubin ≤2ULN（or for subjects with Gilbert's syndrome or lymphoma invading the liver < 3 ULN）；
   4. Baseline oxygen saturation > 92% on room air；
   5. Left ventricular ejection fraction (LVEF) ≥50% assessed by echocardiography or radionuclide activity angiography (MUGA) within 1 month of enrollment；
7. Adequate vascular access for leukapheresis procedure;
8. Women of childbearing potential must agree to use highly effective methods of contraception for at least 28 days prior to lymphocyte clearance chemotherapy through 1 year after Relmacabtagene Autoleucel infusion; Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 1 year after Relmacabtagene Autoleucel infusion.

Exclusion Criteria:

1. Lymphoma involving the central nervous system (CNS)；
2. History of another primary malignancy that has not been in remission for at least 2 years;
3. History of Richter's transformation of chronic lymphocytic leukemia or primary mediastinal B-cell lymphoma；
4. Subjects has HBV, HCV, HIV or syphilis infection at the time of screening;
5. Deep venous thrombosis (DVT)/Pulmonary embolism (PE), or DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
6. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection;
7. Presence of acute or chronic graft-versus-host disease (GVHD);
8. History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
9. Pregnant or nursing women;
10. Subjects Received an autologous or allogeneic hematopoietic stem cell transplant；
11. Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
12. Received CAR T-cell or other genetically-modified T-cell therapy previously；
13. Received live vaccination within 6 weeks prior to lymphocyte clearance chemotherapy；
14. History of severe hypersensitivity reactions to any of the drug ingredients used in this study product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate Per the Lugano Classification as Determined by Study Investigators | up to 2 years after Relmacabtagene Autoleucel infusion
  Complete Response Rate (CRR): percentage of participants with CR [complete metabolic response (CMR); complete radiological response (CRR)]. CMR: positron emission tomography (PET) 5-point scale (5-PS) scores of 1 (no uptake above background), 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass); no new lesions; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow (BM). CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter of lesion (LDi); no extralymphatic sites of disease; absent non-measured lesion (NMLs); organ enlargement regress to normal; no new sites; and bone marrow normal by morphology.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per the Lugano Classification as Determined by Study Investigators | up to 2 years after Relmacabtagene Autoleucel infusion
  ORR: percentage of participants with CR [CMR;CRR] or PR [partial metabolic response (PMR); partial radiologic response (PRR)].CMR: PET 5PS scores of 1 (no uptake above background, 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass; no new lesions; no evidence of FDG-avid disease in BM. CRR:target nodes/nodal masses regressed to ≤ 1.5 cm in LDi;no extralymphatic sites of disease;absent NMLs;organ enlargement regress to normal;no new sites;bone marrow morphology normal. PMR:scores 4 (uptake moderately > liver),5 (uptake markedly > liver, new lesions) with reduced uptake compared with baseline and residual mass;no new lesions;responding disease at interim/residual disease at end of treatment (EOT).PRR: ≥ 50% decrease in sum of the product of perpendicular diameters (SPD) of up to 6 target measurable nodes and extra-nodal sites;absent/normal, regressed, but no increase of NMLs;spleen regressed by > 50% in length beyond normal;no new sites.
Duration of Response (DOR) Per the Lugano Classification | up to 2 years after Relmacabtagene Autoleucel infusion
  DOR is defined only for participants who experience an objective response after Relmacabtagene Autoleucel infusion and is the time from the first objective response to disease progression or death from any cause. Objective response is defined in outcome measure (OM) 2.
Event-Free Survival (EFS) | up to 2 years after Relmacabtagene Autoleucel infusion
  First infusion date of Relmacabtagene Autoleucel to data cut off
Progression-Free Survival (PFS) | up to 2 years after Relmacabtagene Autoleucel infusion
  PFS is defined as the time from the Relmacabtagene Autoleucel infusion date to the date of disease progression per Lugano classification or death from any cause.
Overall Survival (OS) | up to 2 years after Relmacabtagene Autoleucel infusion
  OS is defined as the time from Relmacabtagene Autoleucel infusion to the date of death from any cause.
Types, frequency, and severity of adverse events and laboratory anomalies | up to 2 years after Relmacabtagene Autoleucel infusion
  Physiological parameter
Pharmacokinetic (PK)- Cmax of Relmacabtagene Autoleucel | up to 1 year after Relmacabtagene Autoleucel infusion
  Maximum observed concentration of Relmacabtagene Autoleucel in peripheral blood
Pharmacokinetic (PK)- Tmax of Relmacabtagene Autoleucel | up to 1 year after Relmacabtagene Autoleucel infusion
  Time to maximum concentration of Relmacabtagene Autoleucel in peripheral blood
Pharmacokinetic (PK)- AUC of Relmacabtagene Autoleucel | up to 1 year after Relmacabtagene Autoleucel infusion
  Area under the concentration vs time curve of Relmacabtagene Autoleucel
The concentration of Car-T cell | up to 1 year after Relmacabtagene Autoleucel infusion
  The concentration of Car-T cell in peripheral blood
The change of serum cytokines concentration | up to 1 year after Relmacabtagene Autoleucel infusion
  The change of serum cytokines(IL-2、IL-4、IL-6、IL-8、IL-10、IL-17A、IFN-γ、TNF-α、IFN-α) concentration after Relmacabtagene Autoleucel infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No